CLINICAL TRIAL: NCT04949581
Title: Effect Of Bioelectric Therapy On Sternal Instability In Patients With Median Sternotomy After Heart Valve Surgery: A Randomized Clinical Trial
Brief Title: Effect Of Bioelectric Therapy On Sternal Instability In Patients With Median Sternotomy After Heart Valve Surgery
Acronym: SI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Al Shaymaa Shaaban Abd El Azeim, al shaymaa shaaban abd el azeim, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: p.t.REC/012/003250
Record Dates: First submitted 2021-06-25; First posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Heart Valve Surgery
Keywords: bioelectric therapy; median sternotomy; heart valve surgery

STUDY DESIGN:
Intervention Model Description: bioelectric therapy and routine cardiac rehabilitation program
Who Masked: Participant, Outcomes Assessor
Masking Description: random generator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bioelectric therapy (Experimental): patients will receive micro-current electrical stimulation three times/week for four weeks
  Interventions: Other: bioelectric therapy; Other: cardiac rehabilitation program
- cardiac rehabilitation programe (Active Comparator): patients will receive a cardiac rehabilitation program three times/week for four weeks
  Interventions: Other: cardiac rehabilitation program

INTERVENTIONS:
Other: bioelectric therapy — the patient will receive microcurrent therapy from a supine lying position. the negative electrode on the incision area and the positive electrode proximal. the intensity will be less than 20 microamperes and frequency at 20 HZ.
  Arms: bioelectric therapy
Other: cardiac rehabilitation program — the patient will receive cardiac rehabilitation program

SUMMARY:
The aim of this study is to investigate the effect of bioelectric therapy on sternal instability in patients with median sternotomy after heart valve surgery.

DETAILED DESCRIPTION:
Valvular heart disease constitutes a growing healthcare problem with a general prevalence of 2%-5% and a prevalence of 13% after the age of 75 years Heart valve surgery can be a lifesaving procedure for patients with severe symptomatic heart valve disease. Nevertheless, following the surgery, up to 27% of patients may require readmission within 30 days after discharge. Following heart valve surgery, some patients report anxiety and worries related to readmission and reoperations, postoperative complications, and deconditioning which may prevent or delay return to work and limit activities of daily living.Over the past 30 years, bone-growth stimulators have become a critical component in fracture care. They can be classified into four categories: direct-current (DC) devices, inductive coupling, noninvasive capacitive coupling, and low-intensity ultrasound. Microcurrent electrical stimulation ( MES) is the therapeutic use of constant (DC) and pulsed (interrupted) currents, where the stimulus amplitude is in the micro amperage (millionth of an ampere) range. MES is defined as those of less than 1 mA or 1000 μ, (MES < 1 mA). This form of electrical stimulation tends to be applied at the suspensory or very low sensory level and they are not designed to stimulate muscle contraction. Generators that produce MES were originally called microcurrent electrical neuromuscular stimulators (MENS). However, the stimulation pathway is not the usual neural pathway, and they are not designed to stimulate muscle contraction. Consequently, this type of generator was subsequently referred to as a microcurrent electrical stimulator (MES). The use of MES may be an adjunctive modality in the treatment of fractures or injury sites, especially fractures prone to nonunion. Fracture healing may be accelerated by passing a monophasic current through the fracture site. Getting the current into the bony area without an invasive technique is difficult.forty subjects will be allocated to two groups; one group will receive micro-current therapy and routine cardiac rehabilitation program both for four weeks and the control group will receive the cardiac rehabilitation program only for four weeks.

ELIGIBILITY:
Inclusion Criteria:

1. there age between 40 and 50 years,
2. hemodynamic stability
3. BMI from 25 to 29.9 kg/m2,
4. they will have acute sternal instability.

Exclusion Criteria:

1. previous thoracic surgery
2. elective and urgent coronary artery bypass surgery
3. respiratory insufficiency after surgery manifesting hypoxemia with partial pressure of oxygen in arterial blood <60 mmHg
4. renal insufficiency with serum creatinine ≥1.8 mg/dl after surgery
5. low cardiac output syndrome with ST segment elevation in multiple electrocardiogram leads, cardiac arrhythmias, or hypotension, according to the American College of Cardiology Foundation and American Heart Association

Ages: 40 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-07-15 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
sternal instability | up to four weeks
  sternal instability scale will be used for assessment. this scale has four points. zero mean more stability and three mean completly separated

SECONDARY OUTCOMES:
sternal separation | up to four weeks
  ultrasound unit will be used for assessing the separation between sternum edges